CLINICAL TRIAL: NCT06523803
Title: A Phase 1, Open-label, Multicenter Study of ZW171 in Participants With Advanced or Metastatic Ovarian Cancer, Non-small Cell Lung Cancer (NSCLC), and Other Mesothelin Expressing Cancers
Brief Title: A Study of ZW171 in Participants With Advanced or Metastatic Mesothelin-expressing Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Zymeworks BC Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZWI-ZW171-101; 2024-511119-11 (EudraCT Number)
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Mesothelin-expressing Advanced Cancers
Keywords: Advanced or Metastatic Cancers; ADC; Antibody drug conjugate
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZW171 (Experimental)
  Interventions: Drug: ZW171

INTERVENTIONS:
Drug: ZW171 — Administered per protocol requirements

SUMMARY:
This study is being done to find out if ZW171 is safe and can treat participants with advanced (locally advanced [inoperable] and/or metastatic) mesothelin-expressing cancers.

DETAILED DESCRIPTION:
Part 1 of the study will evaluate the safety and tolerability of ZW171. Part 2 of the study will evaluate the anti-tumor activity of ZW171 while continuing to evaluate the safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of cancers with evidence of locally advanced (unresectable) and/or metastatic disease. Cancers that are refractory to all available standard of care (SOC) treatment, cancers for which no SOC treatment is available, or the participant cannot tolerate or refuses SOC therapy.
* An Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
* Adequate cardiac left ventricular function, as defined by left ventricular ejection fraction ≥ 50% as determined by either echocardiogram or multigated acquisition scan.
* Adequate organ function.

Exclusion Criteria:

* Known additional malignancy that is progressing or that has required active treatment.
* Undergone prior allogenic tissue (e.g., hematopoietic stem cell) or solid organ transplantation within the last 5 years.
* Ongoing, clinically significant toxicity (Grade ≥ 2) associated with prior cancer therapies, with the exception of alopecia.
* Advanced/metastatic, symptomatic, visceral spread, at risk of life-threatening complications in the short-term (including participants with massive uncontrolled effusion [pleural, pericardial], pulmonary lymphangitis, active unresolved bowel obstruction, massive ascites [requiring paracentesis >2 times within 2 weeks prior to the first dose], and over 50% liver involvement).
* Acute or chronic uncontrolled renal disease, pancreatitis, or liver disease (with exception of participants with Gilbert's Syndrome, asymptomatic gall stones, liver metastases, or stable chronic liver disease per investigator assessment).
* Active or recurrent clinically significant autoimmune disease requiring systemic high-dose corticosteroids or immunosuppressive drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs; Part 1) | Up to 3 weeks
  Number of participants who experienced a DLT. DLTs include specifically defined adverse events (AEs) considered to be related to ZW171
Incidence of adverse events (AEs; Parts 1 and 2) | Up to approximately 2 years
  Number of participants who experienced AEs or serious adverse events (SAEs)
Incidence of cytokine release syndrome (CRS; Parts 1 and 2) | Up to approximately 2 years
  Number of participants who experienced CRS
Incidence of neurotoxicity, including immune effector cell-associated neurotoxicity syndrome (ICANS; Parts 1 and 2) | Up to approximately 2 years
  Number of participants who experienced neurotoxicity, including ICANS
Incidence of clinical laboratory abnormalities (Parts 1 and 2) | Up to approximately 2 years
  Number of participants who experienced a maximum severity of Grade 3 or higher post-baseline laboratory abnormality, including either hematology or chemistry. Grades are defined using National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
Confirmed objective response rate (Part 2) | Up to approximately 2 years
  Number of participants who achieved a best overall response of either confirmed complete response (CR) or partial response (PR) during treatment according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Confirmed objective response rate (Part 1) | Up to approximately 2 years
  Number of participants who achieved a best overall response of either confirmed CR or PR during treatment according to RECIST v1.1
Duration of response (DOR; Part 2) | Up to approximately 2 years
  The time from the first objective response (CR or PR) to the first documented progressive disease (PD) per RECIST v1.1 or death within 30 days of last dose of study treatment from any cause. Only participants who achieve a confirmed response will be included in the analysis
Progression-free survival (PFS), including 1-year PFS (Part 2) | Up to approximately 2 years
  The time from the first dose of study treatment to the date of first documented PD per RECIST v1.1 or death from any cause
Disease control rate (DCR; Part 2) | Up to approximately 2 years
  Number of participants who achieved a best response of CR, PR, non-CR/non-PD (for participants who have only non-target lesions), or stable disease (SD) during treatment per RECIST v1.1
Overall survival (OS), including 1-year OS (Part 2) | Up to approximately 2 years
  The time from the first dose of ZW171 until the date of death from any cause
Serum concentration of ZW171 (Parts 1 and 2) | Up to approximately 7 months
  Maximum serum concentration and trough concentration of ZW171
Incidence of anti-drug antibodies (ADAs; Parts 1 and 2) | Up to approximately 7 months
  Number of participants who develop ADAs

CONTACTS AND LOCATIONS:
Overall Officials: Pranshul Chauhan, MSc, MB, BCh, BAO, Study Director — Zymeworks BC Inc.
Locations (15):
- United States (7):
  - University of Southern California - Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Norton Cancer Institute, Louisville, Kentucky
  - Icahn School of Medicine at Mount Sinai (ISMMS) - The Blavatnik Family-Chelsea Medical Center, New York, New York
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Washington, Seattle, Washington
- Universitaetsklinikum Dresden, Dresden, Germany
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Marys Hospital, Seoul
- United Kingdom (3):
  - Guys and St Thomas' NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No